CLINICAL TRIAL: NCT01224197
Title: Phase I, Open Label, Randomized Study to Examine the Pharmacokinetics, Safety and Tolerability of Different Oral Doses of TMC435 After Single and Repeated Dosing in Healthy Chinese Subjects
Brief Title: TMC435 HPC1004 - Phase I Study Investigating the Pharmacokinetics of TMC435 in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017482
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis C
Keywords: TMC435HPC1004; TMC435; HCV; Hepatitis C; Healthy Chinese volunteer
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): TMC435 100 or 200 mg capsule one single dose
  Interventions: Drug: TMC435
- 002 (Experimental): TMC435 100 or 200 mg capsule once daily for 5 days
  Interventions: Drug: TMC435

INTERVENTIONS:
Drug: TMC435 — 100 or 200 mg capsule, one single dose
  Arms: 001
Drug: TMC435 — 100 or 200 mg capsule, once daily for 5 days
  Arms: 002

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, safety and tolerability of single and multiple oral doses of TMC435 in Chinese healthy volunteers. Pharmacokinetics (PK) means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body.

DETAILED DESCRIPTION:
TMC435 is being investigated for the treatment of chronic hepatitic C infection. The results of this study will provide dosing recommendations for the administration of TMC435 in Chinese HCV-infected patients. This is a Phase I, open label (both participant and investigator know the name of the medication given at certain moment), randomized (study medication is assigned by chance) study to investigate the pharmacokinetics, safety and tolerability of TMC435 after single and repeated intakes. Each participant will receive 2 treatments. First, participants will receive TMC435 as a single dose of 100 or 200 mg. Thereafter, in the multiple dose part, 100 or 200 mg TMC435 will be administered during 5 consecutuve days every morning. Both treatments will be administered with food. There will be a washout period of at least 72 hours between the 2 treatments. The main focus of the trial is the pharmacokinetic characteristics (level-profile of TMC435 over time in the blood stream). This evaluation requires multiple blood samples from Day 1 till Day 3 in the first session and from Day 1 till Day 11 in the second session. Safety assessments (blood and urine tests, blood pressure, pulse, electrocardiogram, and physical examination) will follow a different schedule and will be performed during each treatment period, up to 4 weeks after the last. Each volunteer participate in 2 treatments, i.e., single dose period and multiple dose period. In the single dose part, planned doses will be 100 or 200 mg TMC435. In the multiple dose part, TMC435 will be administered during 5 consecutive days every morning.

ELIGIBILITY:
Inclusion Criteria:

* Healthy based on a medical evaluation including medical history, physical examination, blood tests and electrocardiogram. Body Mass Index of 18.0 to 30.0 kg/m² and non-smoker or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months.

Exclusion Criteria:

* Infection with Hepatitis A, B or C virus
* infection with the Human Immunodeficiency Virus (HIV)
* Women who are pregnant or breastfeeding
* History of, or any current medical condition which could impact the safety of the participant in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
plasma concentration of TMC435 after a single oral dose of 100 and 200 mg TMC435 in healthy Chinese volunteers in fed conditions | measured on Day 1, 2, 3
plasma concentration of TMC435 after a multiple oral dose of 100 and 200 mg TMC435 in healthy Chinese volunteers in fed conditions | measured on Day 4 until 11

SECONDARY OUTCOMES:
Safety and tolerability of TMC435 after single oral dose of 100 and 200 mg in healthy Chinese volunteers | Day 1 until Day 3
Safety and tolerability of TMC435 after multiple oral dose of 100 and 200 mg q.d. for 5 days in healthy Chinese volunteers | Day 4 until Day 11 and 12 to 15 days and 38 to 43 days after last intake as safety follow up

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (1):
- Shatin, Hong Kong